CLINICAL TRIAL: NCT02941172
Title: Cannabinoid CB1 Receptors in Human Brown Adipose Tissue
Brief Title: CB1 Receptors in Human Brown Adipose Tissue
Acronym: CANBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, Professor, Turku University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 42/2014
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: Brown adipose tissue; Cannabinoid receptor; PET imaging; Metabolism
MeSH Terms: conditions — Obesity | interventions — 5-((3-fluoromethoxy)phenyl)-3-(1-phenylethylamino)-1-(4-trifluoromethylphenyl)pyrrolidin-2-one; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- [18F]FMPEP-d2 in warm conditions (Other): PET scan is performed using PET radiotracer [18F]FMPEP-d2 in standard room temperature conditions.
  Interventions: Other: [18F]FMPEP-d2
- [18F]FMPEP-d2 in cold conditions (Other): PET scan is performed using PET radiotracer [18F]FMPEP-d2 during controlled cold exposure.
  Interventions: Other: Cold exposure; Other: [18F]FMPEP-d2
- [18F]FDG in cold conditions (Other): PET scan is performed using PET radiotracer [18F]FDG during controlled cold exposure.
  Interventions: Other: Cold exposure; Other: [18F]FDG

INTERVENTIONS:
Other: Cold exposure — Controlled cold exposure is performed before and during PET scan
  Arms: [18F]FDG in cold conditions; [18F]FMPEP-d2 in cold conditions
Other: [18F]FMPEP-d2 — PET radiotracer used in imaging
  Arms: [18F]FMPEP-d2 in cold conditions; [18F]FMPEP-d2 in warm conditions
Other: [18F]FDG — PET radiotracer used in imaging
  Arms: [18F]FDG in cold conditions

SUMMARY:
This study investigates cannabinoid CB1 receptors in human brown adipose tissue (BAT) and other tissues using positron emission tomography (PET) imaging. Subjects will be scanned in room temperature conditions and during controlled cold exposure, and the density of CB1 receptors in BAT and other tissues will be quantified. The investigators hypothesize, that cannabinoid signaling is increased in cold conditions, when BAT is metabolically active.

Understanding the mechanisms of BAT activation and the role of endocannabinoids in humans is important and beneficial in fighting against the epidemic of obesity and diabetes.

DETAILED DESCRIPTION:
Endocannabinoids have an important role in regulating energy balance and metabolism. Cannabinoid 1 receptors (CB1) are found in several tissues such as brown adipose tissue (BAT). Endocannabinoids and CB1 receptors participate in the control of lipid and glucose metabolism, and blockage of CB1 receptors has been found to improve metabolic factors linked to obesity and cardiovascular disease, making CB1 antagonists potential drugs against obesity and diabetes.

In this study the investigators use a PET radiotracer [18F]FMPEP-d2, which binds to CB1 receptors in vivo, to quantify the CB1 receptor density in BAT, white adipose tissue, muscle and the brain. This study is done once in warm conditions and once during controlled cold exposure. To verify whether the subject has metabolically active BAT, an additional PET scan with the radiotracer [18F]FDG is performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Group 1: BMI 20-26 kg/m2, Group2: BMI 27-40 kg/m2

Exclusion Criteria:

* BMI < 20 kg/m2or BMI > 40 kg/m2
* Any chronic disease that could affect the study outcome, including medicated type 2 diabetes
* Mental disorder or poor compliance
* Eating disorder or excessive use of alcohol, tobacco smoking or drug use
* Past dose of radiation
* Presence of any ferromagnetic objects that would make MR imaging contraindicated
* Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
CB1 density of brown adipose tissue acquired with PET | within one study day
  PET imaging is used to quantify CB1 receptors in tissues

SECONDARY OUTCOMES:
Glucose uptake of brown adipose tissue acquired with PET | within one study day
  PET imaging is used to quantify glucose uptake in tissues

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, M.D., Ph.D., Principal Investigator — Turku PET Centre (Turku University Hospital)
Locations (1):
- Turku PET Centre (Turku University Hospital), Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lahesmaa M, Eriksson O, Gnad T, Oikonen V, Bucci M, Hirvonen J, Koskensalo K, Teuho J, Niemi T, Taittonen M, Lahdenpohja S, U Din M, Haaparanta-Solin M, Pfeifer A, Virtanen KA, Nuutila P. Cannabinoid Type 1 Receptors Are Upregulated During Acute Activation of Brown Adipose Tissue. Diabetes. 2018 Jul;67(7):1226-1236. doi: 10.2337/db17-1366. Epub 2018 Apr 12. PMID 29650773